CLINICAL TRIAL: NCT04359758
Title: Streamlined Genetic Testing in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marc D Schwartz, Professor of Oncology, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00001073; P30CA051008 (NIH)
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proactive Streamlined Genetic Education and Testing (Experimental): Participants randomized to this arm will proactively receive genetic education print materials and the option to proceed directly with genetic testing.
  Interventions: Behavioral: Proactive Streamlined Genetic Education and Testing
- Usual Care (Active Comparator): Participants in this arm will be sent a referral letter recommending that they schedule a genetic counseling session and providing them with contact information to do so.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Proactive Streamlined Genetic Education and Testing — This intervention consists of the proactive delivery of genetic education print materials followed by streamlined and facilitated access to genetic testing.
  Arms: Proactive Streamlined Genetic Education and Testing
Behavioral: Usual Care — This intervention consists of a standard genetic referral letter that notified the participant that he qualified for genetic referral, recommends the scheduling of a genetic counseling session and provides a telephone number for scheduling.
  Arms: Usual Care

SUMMARY:
The goal of this pilot randomized controlled trial is to evaluate the impact and efficacy of a streamlined genetic education and testing intervention for men with prostate cancer. Eligible men are prostate cancer survivors who meet criteria for genetic counseling referral. After completing a baseline survey, participants (n=120) are randomized to Streamlined Genetic Testing (ST) or Usual Care (UC). Participants in ST are able to review genetic education materials and then proceed directly to genetic testing. Participants in UC will be provided with a referral for standard individual genetic counseling. Two months after randomization all participants will be contacted to complete a follow-up survey.

DETAILED DESCRIPTION:
Genetic testing is part of clinical care for women with breast and ovarian cancer. Guidelines have led to increasing genetic testing participation among eligible women. Identifying pathogenic variants (PVs) in cancer susceptibility genes has important treatment, management and risk reduction implications for patients and their family members. Men are just as likely as women to carry a PV in a cancer risk gene and men with prostate cancer are at particularly high risk for carrying a PV. NCCN guidelines recommend germline genetic testing in men with metastatic prostate cancer or with Gleason 7+ prostate cancer. These guidelines are likely to expand given recent studies suggesting that 17% of prostate cancer patients may harbor a cancer susceptibility PV and that current referral criteria miss many of these patients. Prostate cancer patients with a PV in BRCA1 or BRCA2 (BRCA) have more aggressive prostate cancers, are at risk for other primary cancers (e.g., male breast and pancreatic) and their family members are at risk for a variety of cancers. Thus, genetic testing of prostate cancer patients has implications for treatment, management, and risk reduction for the patient and his family members.

Despite these benefits and existing referral guidelines, few men with prostate cancer are tested. This reflects low genetic counseling referral and participation, since men who attend genetic counseling get tested at the same high rate as women. Low participation is likely due to underestimation of the personal health relevance of testing and lack of physician genetic counseling referral. Thus, the requirement to obtain individual genetic counseling prior to genetic testing may be a barrier to the receipt of guideline consistent genetic testing. Recent evidence suggests that traditional comprehensive, patient-centered, educationally focused pre-test genetic counseling often does not match the needs of patients. Further, as genetic referral guidelines continue to expand, demand for genetic counseling will outstrip delivery capacity. Thus, alternative approaches that raise awareness and facilitate access to genetic testing are needed to maximize our ability to extend the benefits of testing to prostate cancer patients and their family members while at the same time accommodating increased demand and conserving scarce genetic counseling resources.

We will test a proactive and streamlined pre-test genetic education (ST) print intervention designed to speed, simplify and target genetic testing delivery for prostate cancer patients. Participants randomized to ST will have the option to proceed directly to genetic testing bypassing traditional pre-test genetic counseling. Usual care (UC) participants will be informed that they meet guidelines for genetic counseling referral and will be provided with contact information to schedule a standard telephone pre-test genetic counseling session. All participants with a PV or variant of uncertain significance (VUS) will be scheduled for a telephone genetic counseling disclosure session. ST participants who are found not to carry a PV or VUS will have this result disclosed via clinical letter while disclosure for all UC participants will be per standard clinical care by the genetic counselor by phone. By proactively identifying eligible patients, providing streamlined information and facilitating genetic testing, the ST intervention will increase awareness, facilitate informed testing decisions, remove the barrier of pre-test genetic counseling and improve genetic testing delivery capacity.

We will enroll eligible prostate patients diagnosed from 2010-2019 who are being followed within radiation and medical oncology clinics at the MedStar Georgetown University Hospital and MedStar Washington Hospital Center. Our specific aims are:

1. Evaluate the impact of ST vs. UC on genetic testing uptake. H1.1: Patients randomized to ST will be more likely to complete genetic testing compared to UC. H1.2: Participants randomized to ST will make better informed genetic testing decisions (characterized by high knowledge, risk comprehension and concordance with attitudes) compared to UC. H1.3: Few patients in the ST arm will opt for traditional genetic counseling prior to testing.
2. Evaluate patient satisfaction and psychosocial outcomes in ST vs. UC. H2.1: Compared to UC, those randomized to ST will be more satisfied with their genetic testing decision and will have less decisional regret.
3. Evaluate the impact of ST vs. UC on uptake of cascade testing in unaffected family members. In exploratory analyses designed to provide effect size estimates, we will compare the arms on rates of genetic testing in relatives of patients found to carry a PV.

Gender and Minorities. Participants will be adult men. Given the racial/ethnic breakdown of the clinics we are recruiting from. We expect that at least 30% of participants will be members of racial/ethnic minority groups.

Recruitment. Working with our clinical collaborators and the Survey, Recruitment and Biospecimen Collection Shared Resource (SRBSR) will obtain contact information of potentially eligible patients from clinical databases and/or the EMR. We will mail an introductory letter describing the study (from the study MPIs and the patient's physician), opt-out postcard/phone number, informed consent document and a print version of the baseline survey to all potentially eligible participants. We will also email electronic versions of these materials. Two-weeks following this mailing, a research assistant (RA) will call patients who have neither opted out nor completed the baseline survey. For men who have not returned the consent document, we will use an IRB-approved verbal consent for completing the baseline survey and request return of the written consent prior to randomization. Following completion of print or electronic consent and the baseline survey, the RA will randomize participants. Men randomized to ST will be sent a priority mail packet with detailed genetic testing educational material. Men randomized to UC will be mailed a letter informing them that they meet guidelines for genetic counseling and provided with contact information to schedule a genetic counseling appointment with a LCCC genetic counselor.

Randomization. Following completion of the baseline survey and consent document, an RA will randomize participants via computer-generated random numbers in blocks of 8 and a ratio of 1:1. Participants will be notified of their random assignment via letter and email.

Assessments. We will administer baseline (T0) a 1- to 2-month (T1) follow-up telephone/electronic surveys. Genetic testing uptake will be assessed via clinical records and basic clinical and demographic information abstracted from the EMR.

Streamlined Testing (ST) Intervention. Men randomized to ST will be sent a priority mail packet with the ST print education materials and information on how to proceed with genetic testing. ST participants will have the option of proceeding directly to genetic testing or scheduling a telephone genetic counseling session. The content of the ST intervention is described in section 5.0 above.

Usual Care (UC). After completion of the baseline survey, UC participants will be sent a letter from their physician indicating that they meet eligibility criteria for genetic testing, recommending that they schedule genetic counseling and providing a contact telephone number to schedule their session. Patients may opt for free telephone genetic counseling.

Genetic Testing. Participants who opt for genetic testing will be offered a standard multigene panel of at least 40 genes, including BRCA and genes associated with potential differential diagnoses (e.g., Lynch syndrome). All testing will be performed by Invitae, a CLIA certified clinical lab not affiliated with the GLCCC. Invitae offers genetic testing free of charge to eligible prostate cancer patients. Prior to proceeding with genetic testing, participants will be required to sign and return a clinical genetic testing consent form, after which we will mail them an at-home DNA kit for saliva collection which will be returned directly to Invitae (shipping costs are pre-paid).

Data Analysis: We will characterize participants by comparing them to decliners on key demographic and clinical variables derived from the EMR. After performing univariate analysis on dependent variables, we will apply any needed normalizing or variance stabilizing transformations. We will follow Consort guidelines for Intent-to-Treat analyses (ITT). We will compare groups at baseline with χ2 and t-tests and will include covariates that are associated with group (p <0.10) in our final models.

Aim 1: Evaluate the impact of Proactive Streamlined Education and Testing (ST) vs. Usual Care (UC) on genetic testing. Analysis: H1.1: Patients randomized to ST will be more likely to complete genetic testing compared to UC. We will use logistic regression to test this hypothesis. After entering significant covariates, we will add intervention arm to test the overall intervention effect. H1.2: Participants randomized to ST will make better informed genetic testing decisions (characterized by high knowledge, risk comprehension and positive attitudes) compared to UC. Using multiple regression, we will enter control/confounding variables and intervention to test the impact of group on our informed decision making outcomes (knowledge, testing attitudes, risk comprehension). H1.3: Few patients in the ST arm will opt for traditional genetic counseling prior to testing. We will conduct descriptive analyses describing the proportion of ST participants who opt for genetic counseling vs. proceed directly to testing vs. opt against testing.

Aim 2: Evaluate patient satisfaction and psychosocial outcomes in ST vs. UC. Analysis: H2.1: Compared to UC, those randomized to ST will be more satisfied with their genetic testing decision and will have less decisional regret. After identifying baseline confounders of each outcome, we will generate linear regression models in which we enter: 1) confounders; 2) genetic test result (dummy coded to generate comparisons of carriers vs. non-carriers and non-carriers vs. untested); 3) group assignment. In the event that we have an insufficient number of PV carriers for these analyses, we will categorize test result into two levels (tested vs. untested) and evaluate results among PV carriers more descriptively. Results of Aim 2 analyses will be primarily focused on generating effect size estimates for our planned trial of newly diagnosed prostate cancer patients.

Aim 3: Evaluate the impact of ST vs. UC on uptake of cascade testing in unaffected family members. In exploratory analyses designed to provide effect size estimates for our planned R01, we will use t-test to compare the ST to UC on the number of relatives of PV carriers who undergo cascade genetic testing.

Power: Power estimates are for 2-tailed tests (α=.05). The study is powered based on our primary outcome of patient genetic testing uptake. We expect no attrition since data will be abstracted from clinic records. We will enroll 120 participants in order to attain 80% power to detect a clinically meaningful increase of 25% in test uptake from 20% in UC to 45% in ST. For secondary outcomes, assuming 10% attrition, we will have 80% power to detect modest effect sizes of d=.54 SDs.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Diagnosed with metastatic prostate cancer or Gleason 7+ prostate cancer
* Diagnosed between 2010-2020

Exclusion Criteria:

* Age 81 or older
* Previous cancer genetic counseling or testing
* Previously scheduled for cancer genetic counseling or testing
* Cannot participate in English
* Are not capable of providing informed consent

Ages: 21 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University Medical Center/Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with Georgetown University.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: 12-36 months after publication.
Access Criteria: Investigator who proposes to use the data must obtain approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and execute a data use/sharing agreement with Georgetown University.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potentially eligible participants were identified via the electronic health record at Medstar Georgetown University Hospital. The first participant was enrolled in February 2020 and the last participant was enrolled in March 2021.
Pre-assignment Details: Of 216 potentially eligible participants, 112 completed the baseline survey and were randomized. Five participants were found to be ineligible after randomization (i.e., protocol violation). Thus, the final sample was comprised of 107 men who were randomized to ST (n=53) vs UC (n=54).
Period: Overall Study
Arm/Group | Proactive Streamlined Genetic Education and Testing | Usual Care
Started | 56 | 56
Completed | 53 | 54
Not Completed | 3 | 2
Not completed — Protocol Violation | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proactive Streamlined Genetic Education and Testing | Usual Care | Total
Number analyzed (Participants) | 53 | 54 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (7.4) | 71.6 (7.0) | 71.2 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 53 | 54 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 51 | 52 | 103
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 15 | 28
  White | 37 | 38 | 75
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 53 | 54 | 107
Education [Count of Participants; unit: Participants]
  College Degree | 24 | 34 | 58
  Less Than College Degree | 29 | 20 | 49
Marital Status [Count of Participants; unit: Participants]
  Married/Partnered | 40 | 39 | 79
  Not Married/Partnered | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completing Genetic Testing
Description: Receipt of genetic testing results as indicated in clinic records
Time Frame: Three Months Post-Randomization
Population: Intent to Treat (all participants assigned to ST or UC).
Measure: Count of Participants; unit: Participants
Arm/Group | Proactive Streamlined Genetic Education and Testing | Usual Care
Number analyzed (Participants) | 53 | 54
Participants
  Completed Genetic Testing | 22 | 15
  Declined Genetic Testing | 31 | 39
Statistical Analysis 1: Comparison: Proactive Streamlined Genetic Education and Testing vs Usual Care; The study was powered assuming 10% genetic testing uptake UC compared to 35% in ST. assuming these uptake rates and a two-tailed alpha of 0.05, a sample size of n=50 per arm would yield greater than 80% power; Test type: Superiority; p = 0.14, Chi-squared
Statistical Analysis 2: Comparison: Proactive Streamlined Genetic Education and Testing vs Usual Care; Because education and marital status have been associated with genetic testing participation in prior research, we conducted a follow-up analysis in which we adjusted for education and marital status; Test type: Superiority; p = 0.039, Regression, Logistic; Odds Ratio (OR) = 2.57, 95% CI 2-sided [1.05 to 6.29]

2. Secondary Outcome: Decision Satisfaction
Description: Satisfaction with Decision Scale Higher values indicate greater satisfaction with the genetic testing decision. Range = 6 to 30.
Time Frame: 3 Months Post Randomization
Population: Participants completing the 3-month follow-up assessment. Three participants who completed the 3-month follow-up failed to complete this scale. Thus, the final sample size for this analysis was N=103.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Proactive Streamlined Genetic Education and Testing | Usual Care
Number analyzed (Participants) | 52 | 51
score on a scale | 21.3 (6.6) | 23.2 (5.1)
Statistical Analysis 1: Comparison: Proactive Streamlined Genetic Education and Testing vs Usual Care; Test type: Superiority; p = 0.13, t-test, 2 sided; 101 degrees of freedom

3. Secondary Outcome: Decisional Regret
Description: Decision Regret Scale Higher score indicates greater regret regarding the genetic testing decision Range = 0 to 100
Time Frame: 3 Months Post Randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Proactive Streamlined Genetic Education and Testing | Usual Care
Number analyzed (Participants) | 53 | 51
score on a scale | 26.5 (21.4) | 25.4 (18.6)
Statistical Analysis 1: Comparison: Proactive Streamlined Genetic Education and Testing vs Usual Care; Test type: Superiority; p = 0.78, t-test, 2 sided; df=102

4. Secondary Outcome: Distress
Description: Patient Reported Outcomes Measurement Information System - Depression Short Scale 6A T-Scores (Mean = 50 and SD = 10; Range = 38.4 to 80.3) Higher scores indicate greater depression
  Patient Reported Outcomes Measurement Information System - Anxiety Short Scale 6A T-Scores (Mean = 50, SD = 10; Range = 39.1 to 82.7) Higher scores indicate more anxiety
Time Frame: 3 Months Post Randomization
Population: Total number of randomized participants who completed the PROMIS depression and anxiety measures
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Proactive Streamlined Genetic Education and Testing | Usual Care
Number analyzed (Participants) | 52 | 52
T-Score
  Anxiety - Baseline | 48.5 (8.5) | 48.4 (9.1)
  Anxiety - 3-Months | 47.5 (9.2) | 47.4 (8.8)
  Depression - Baseline | 43.6 (6.8) | 47.4 (8.7)
  Depression - 3-Months | 44.0 (7.8) | 45.9 (8.6)
Statistical Analysis 1: Comparison: Proactive Streamlined Genetic Education and Testing vs Usual Care; Analysis of PROMIS anxiety; Test type: Superiority; p = 0.97, ANCOVA; df = 1, 101
Statistical Analysis 2: Comparison: Proactive Streamlined Genetic Education and Testing vs Usual Care; Analysis of PROMIS Depression; Test type: Superiority; p = 0.34, ANCOVA; df = 1, 101

ADVERSE EVENTS:
Time Frame: 3-Months
Arm/Group | Proactive Streamlined Genetic Education and Testing | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/55
Other Adverse Events (participants affected / at risk) | 0/53 | 0/55

LIMITATIONS AND CAVEATS:
Small sample size due to the the fact that this was a pilot trial. This impacted statistical power and ability to conduct subgroup analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT04359758/Prot_SAP_000.pdf